CLINICAL TRIAL: NCT00000520
Title: Prevention of Coronary Aneurysms in Kawasaki Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 39; R01HL034545 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Coronary Aneurysm; Heart Diseases; Mucocutaneous Lymph Node Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Aneurysm; Heart Diseases; Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulins, Intravenous; Aspirin

INTERVENTIONS:
Drug: immunoglobulins, intravenous
Drug: aspirin

SUMMARY:
To test the efficacy of intravenous gamma globulin (IVGG) in preventing coronary artery aneurysms in children with Kawasaki Syndrome.

DETAILED DESCRIPTION:
BACKGROUND:

Kawasaki Syndrome is an acute febrile illness that occurs predominantly in previously healthy young children. It is of unknown etiology and was first described in Japan in 1967. The illness carries an acute mortality rate of approximately 3 percent. The Centers for Disease Control defines Kawasaki Syndrome as a fever lasting five or more days for which no explanation can be found. Patients also must have at least four of the following symptoms: bilateral conjunctival infection; infected or fissured lips, pharynx, or a 'strawberry tongue'; erythema of the palms or soles, or edema of the hands or feet, or generalized or periungual desquamation; rash; and cervical lymphadenopathy.

Coronary artery aneurysms occur in 15-20 percent of children with the illness. In the past, no treatment had been shown to be effective in preventing this complication. Investigators in Japan began to use IVGG to reduce the aneurysm formation. Preliminary results showing the usefulness of this therapy led to a multicenter trial in Japan in which 400 mg/kg/day of IVGG were given for five days to children also receiving aspirin for the condition. Results of the Japanese trial showed that within 29 days of the onset of the disease, coronary artery dilatation had developed in 42 percent of the aspirin-treated children and in 15 percent of the IVGG and aspirin-treated children.

DESIGN NARRATIVE:

Phase I was randomized, unblinded and stratified by age, sex, and center. Subjects were randomized to receive either 80 to 120 mg/kg/day of aspirin through day 14 of illness, subsequently reduced to 3 to 5 mg/kg/day as a single daily dose or to 400 mg/kg/day of intravenous gamma globulin for four consecutive days plus aspirin as above. Primary endpoint was formation of aneurysms as demonstrated by echocardiograms. Follow-up was for 7 weeks.

Phase II of the trial began enrollment of 549 patients in May 1986 and ended enrollment in November 1989. Two hundred and seventy six children were randomized to receive 400 mg/kg of intravenous gamma globulin over four consecutive days. Two hundred and seventy-three received a single infusion of 2 g/kg of body weight over 10 hours. Both treatment groups received 100 mg/kg of aspirin per day through day 14 and then 3 to 5 mg/kg per day. The primary outcome variables were the presence or absence of coronary artery abnormalities evident at the two week and seven week follow-up examinations. Echocardiograms were obtained for 523 children at the two week visit and for 520 children at the seven week visit.

ELIGIBILITY:
Boys and girls who met the CDC criteria for Kawasaki Syndrome. Subjects were excluded if they presented themselves to the participating centers after the tenth day of illness.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1985-07; Study Completion 1989-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Rosen — Children's Hospital Medical Center, Cincinnati

REFERENCES:
- [Background] Newburger JW, Takahashi M, Burns JC, Beiser AS, Chung KJ, Duffy CE, Glode MP, Mason WH, Reddy V, Sanders SP, et al. The treatment of Kawasaki syndrome with intravenous gamma globulin. N Engl J Med. 1986 Aug 7;315(6):341-7. doi: 10.1056/NEJM198608073150601. PMID 2426590
- [Background] Burns JC, Geha RS, Schneeberger EE, Newburger JW, Rosen FS, Glezen LS, Huang AS, Natale J, Leung DY. Polymerase activity in lymphocyte culture supernatants from patients with Kawasaki disease. Nature. 1986 Oct 30-Nov 5;323(6091):814-6. doi: 10.1038/323814a0. PMID 2430187
- [Background] Shulman ST, Rowley AH. Does Kawasaki disease have a retroviral aetiology? Lancet. 1986 Sep 6;2(8506):545-6. doi: 10.1016/s0140-6736(86)90115-7. PMID 2427900
- [Background] Leung DY, Geha RS, Newburger JW, Burns JC, Fiers W, Lapierre LA, Pober JS. Two monokines, interleukin 1 and tumor necrosis factor, render cultured vascular endothelial cells susceptible to lysis by antibodies circulating during Kawasaki syndrome. J Exp Med. 1986 Dec 1;164(6):1958-72. doi: 10.1084/jem.164.6.1958. PMID 3491174
- [Background] Burns JC, Wiggins JW Jr, Toews WH, Newburger JW, Leung DY, Wilson H, Glode MP. Clinical spectrum of Kawasaki disease in infants younger than 6 months of age. J Pediatr. 1986 Nov;109(5):759-63. doi: 10.1016/s0022-3476(86)80689-8. PMID 3772656
- [Background] Gidding SS, Shulman ST, Ilbawi M, Crussi F, Duffy CE. Mucocutaneous lymph node syndrome (Kawasaki disease): delayed aortic and mitral insufficiency secondary to active valvulitis. J Am Coll Cardiol. 1986 Apr;7(4):894-7. doi: 10.1016/s0735-1097(86)80354-0. PMID 3958349
- [Background] Hicks RV, Melish ME. Kawasaki syndrome. Pediatr Clin North Am. 1986 Oct;33(5):1151-75. doi: 10.1016/s0031-3955(16)36113-2. PMID 3532006
- [Background] Melish ME, and Hicks RV. Kawasaki Syndrome. In: John D. Nelson (editor) Current Therapy in Pediatric Infectious Disease, pp. 106-162. The C.V. Mosby Co., 1986.
- [Background] Takahashi M, Mason W, Lewis AB. Regression of coronary aneurysms in patients with Kawasaki syndrome. Circulation. 1987 Feb;75(2):387-94. doi: 10.1161/01.cir.75.2.387. PMID 3802442
- [Background] Leung DY, Burns JC, Newburger JW, Geha RS. Reversal of lymphocyte activation in vivo in the Kawasaki syndrome by intravenous gammaglobulin. J Clin Invest. 1987 Feb;79(2):468-72. doi: 10.1172/JCI112835. PMID 2433307
- [Background] Rowley AH, Gonzalez-Crussi F, Gidding SS, Duffy CE, Shulman ST. Incomplete Kawasaki disease with coronary artery involvement. Prog Clin Biol Res. 1987;250:357-65. No abstract available. PMID 3423049
- [Background] Rowley AH, Shulman ST. The search for the etiology of Kawasaki disease. Pediatr Infect Dis J. 1987 Jun;6(6):506-8. doi: 10.1097/00006454-198706000-00002. No abstract available. PMID 3302905
- [Background] Gidding SS, Duffy CE, Pajcic S, Berdusis K, Shulman ST. Usefulness of echocardiographic evidence of pericardial effusion and mitral regurgitation during the acute stage in predicting development of coronary arterial aneurysms in the late stage of Kawasaki disease. Am J Cardiol. 1987 Jul 1;60(1):76-9. doi: 10.1016/0002-9149(87)90988-x. PMID 3604947
- [Background] Rowley AH, Shulman ST. Kawasaki disease: new etiologic clues and advances in therapy. Pediatr Dermatol. 1987 Aug;4(2):134-5. doi: 10.1111/j.1525-1470.1987.tb00767.x. No abstract available. PMID 3658834
- [Background] Rowley AH, Gonzalez-Crussi F, Gidding SS, Duffy CE, Shulman ST. Incomplete Kawasaki disease with coronary artery involvement. J Pediatr. 1987 Mar;110(3):409-13. doi: 10.1016/s0022-3476(87)80503-6. PMID 3819942
- [Background] Rowley AH, Shulman ST, Preble OT, Poiesz BJ, Ehrlich GD, Sullivan JR. Serum interferon concentrations and retroviral serology in Kawasaki syndrome. Pediatr Infect Dis J. 1988 Sep;7(9):663-6. No abstract available. PMID 3140211
- [Background] Rowley AH, Shulman ST. What is the status of intravenous gamma-globulin for Kawasaki syndrome in the United States and Canada? Pediatr Infect Dis J. 1988 Jul;7(7):463-6. doi: 10.1097/00006454-198807000-00001. No abstract available. PMID 2457202
- [Background] Rowley AH, Duffy CE, Shulman ST. Prevention of giant coronary artery aneurysms in Kawasaki disease by intravenous gamma globulin therapy. J Pediatr. 1988 Aug;113(2):290-4. doi: 10.1016/s0022-3476(88)80267-1. PMID 2456378
- [Background] Leung DY, Cotran RS, Kurt-Jones E, Burns JC, Newburger JW, Pober JS. Endothelial cell activation and high interleukin-1 secretion in the pathogenesis of acute Kawasaki disease. Lancet. 1989 Dec 2;2(8675):1298-302. doi: 10.1016/s0140-6736(89)91910-7. PMID 2480498
- [Background] Newburger JW, Sanders SP, Burns JC, Parness IA, Beiser AS, Colan SD. Left ventricular contractility and function in Kawasaki syndrome. Effect of intravenous gamma-globulin. Circulation. 1989 Jun;79(6):1237-46. doi: 10.1161/01.cir.79.6.1237. PMID 2720925
- [Background] Burns JC, Huang AS, Newburger JW, Reinhart AL, Walsh MM, Hoch S, Leung DY. Characterization of the polymerase activity associated with cultured peripheral blood mononuclear cells from patients with Kawasaki disease. Pediatr Res. 1990 Feb;27(2):109-12. doi: 10.1203/00006450-199002000-00001. PMID 1690383
- [Background] Newburger JW, Takahashi M, Beiser AS, Burns JC, Bastian J, Chung KJ, Colan SD, Duffy CE, Fulton DR, Glode MP, et al. A single intravenous infusion of gamma globulin as compared with four infusions in the treatment of acute Kawasaki syndrome. N Engl J Med. 1991 Jun 6;324(23):1633-9. doi: 10.1056/NEJM199106063242305. PMID 1709446